CLINICAL TRIAL: NCT03960333
Title: Immunometabolism in Pediatric Obesity
Acronym: IPO
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 228816; P20GM109096 (NIH)
Record Dates: First submitted 2019-05-06; First posted 2019-05-23 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Type 2 Diabetes Mellitus; Insulin Resistance
Keywords: Obesity; Type2 Diabetes Mellitus; Type2 Diabetes; Insulin Resistance; Metformin; Pediatric Health
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood, urine, and stool samples may be retained. The blood sample will be used for bioenergetics, immunophenotyping, CD4+ T cell isolations, metabolic control pathway analysis, quantification of plasma CRP, pro-inflammatory, and anti-inflammatory cytokines and adipokines, and analyte analysis. The sample may be used for future research studies on pediatric nutrition. The urine and stool sample will be used for future research studies on pediatric nutrition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Lean: Healthy lean individuals (n=20) defined with a Body Mass Index (BMI) ≥ 5th percentile and <85th percentile for age/sex will be recruited. Participants in this cohort will be asked to complete a one-time study visit.
- Overweight/Obese: Overweight/Obese individuals (n=20) defined with a Body Mass Index (BMI) ≥ 85th percentile for age/sex will be recruited. Participants in this cohort will be asked to complete a one-time study visit.
- Type 2 Diabetes or Insulin Resistant: Obese individuals with Type 2 Diabetes or insulin resistance who have been recently prescribed Metformin and have a Body Mass Index (BMI) ≥ 85th percentile for age/sex (n=20) will be recruited. Participants in this cohort will be asked to complete a two study visits approximately 6 months apart.

SUMMARY:
This is a study to learn about obesity and how insulin resistance and Type 2 Diabetes develops in children.

DETAILED DESCRIPTION:
The main purpose of this proposed study is to determine whether the immunometabolic phenotypes of CD4+T cells from obese children is skewed towards Teff with mTOR-driven glycolysis and away from Tregs with AMPK-driven OXPHOS and whether metformin can reverse the immunometabolic phenotypes.

This study consists of:

1. An observational cross sectional immune and metabolic analysis of several groups of children including lean, overweight/obese, and T2D.
2. A prospective immune and metabolic analysis of newly diagnosed children with T2D or insulin resistance who will be or were recently prescribed metformin as part of their clinical care.

Children with T2D or insulin resistance who will be or were recently prescribed metformin, will be asked to complete two study visits. If completed, the second visit will occur 6 months (+/- 2 weeks) after beginning metformin as part of their clinical care. All other children, will be asked to complete only the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-17 years, inclusive
* Either healthy lean (BMI≥ 5th percentile and <85th percentile for age/sex) or overweight (BMI ≥ 85th percentile and <95th) or obese (BMI ≥ 95th percentile for age/sex)
* For those with BMI≥ 85th percentile for age/sex, parental verbal confirmation that the child had a history of BMI≥ 85th percentile for age/sex for at least six months prior to study enrollment OR
* Age 5 years - 17 years 5 months, inclusive
* Either overweight or obese (BMI≥ 85th percentile for age/sex)
* Parental verbal confirmation that the child had a history of BMI≥ 85th percentile for age/sex for at least six months prior to study enrollment
* Diagnosed with type 2 diabetes mellitus or insulin resistance
* Prescribed metformin (either not yet taking or began taking within 3 weeks of enrollment)

Exclusion Criteria:

* Having an infection (viral, respiratory, gastrointestinal) in the previous 4 weeks
* Genetic or physical conditions impacting mobility over past year as determined by the PI
* Having known chronic illnesses/disorders that may independently affect study outcome measures: type 1 diabetes mellitus, neurologic (e.g. epilepsy), developmental (developmental delay, autism spectrum disorder), endocrine (thyroid, Cushing's), hepatic, autoimmune, cardiac and renal disorders. Also, chronic lung disorders except well controlled asthma that does not require permanent use of inhaled/oral steroids
* Taking any of the following medications that can affect study outcome: antipsychotics, thyroid hormone replacement therapy, inhaled/oral steroids, insulin, anabolic drugs (growth hormone replacement therapy and oxandrolone) and stimulants
* Taking metformin prescribed as part of their clinical care for longer than 3 weeks at the time of enrollment (may begin metformin therapy prescribed as part of their clinical care while enrolled in the study)
* BMI<5th percentile for age/sex (classified as underweight based on CDC growth charts)
* Subjects determined ineligible by the PI or delegated staff.

Ages: 5 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: 110 children ages 5-17 years old will be recruited with the goal that approximately 80 subjects stratified across the following groups will complete the study: i) healthy lean (approximately n=20); ii) overweight/obese (approximately n=40, with the anticipation that approximately 20 of these children will be insulin resistant); iii) overweight/obese with T2D and prescribed Metformin (approximately n=20). Every attempt will be made to ensure that the desired number for each group is achieved and groups are balanced with respect to age, sex and ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
circulating CD4+T cells in Overweight/Obese vs Lean | After completion of all study visits, approximately 2 years.
  We will measure and report the percent of ATP derived from glycolysis and oxidative phosphorylation in circulating CD4+ T cells as well as the % CD4+CD25+CD127lowFoxP3+ cells (Tregs) in overweight/obese vs lean children.
circulating CD4+T cells in Type 2 Diabetic pre/post Metformin | After completion of all study visits, approximately 2 years.
  We will measure and report the percent of ATP derived from glycolysis and oxidative phosphorylation in circulating CD4+ T cells as well as the % CD4+CD25+CD127lowFoxP3+ cells (Tregs) in Type 2 Diabetic children pre and post-Metformin treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Rose, PhD, Principal Investigator — Arkansas Children's Research Institute
Locations (1):
- Arkansas Children's Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The information collected at the study visit, urine, and stool samples, and remaining blood samples may be stored indefinitely and may be used for future research studies on pediatric nutrition or metabolism. Prior to the information collected at the study visit and samples being used for future research studies, the PI will assess the ethics and scientific merit of the proposed research with the samples, and proposed future research will be reviewed by the IRB as may be required.
Supporting Information: CSR
Time Frame: The data and samples will be available after all data has been collected for the study and all samples have been processed for the study. Prior to the information collected at the study visit and samples being used for future research studies, the PI will assess the ethics and scientific merit of the proposed research with the samples, and proposed future research will be reviewed by the Institutional Review Board (IRB) as may be required.
Access Criteria: The samples and health information collected for the study visit may be shared with researchers at the University of Arkansas for Medical Sciences, Arkansas Children's Hospital, or Arkansas Children's Research Institute. The samples may be shared with an outside group. The samples will only have a study number, visit number, and study acronym to maintain confidentiality.

REFERENCES:
- [Result] Rose S, Landes RD, Vyas KK, Delhey L, Blossom S. Regulatory T cells and bioenergetics of peripheral blood mononuclear cells linked to pediatric obesity. Immunometabolism (Cobham). 2024 Apr 25;6(2):e00040. doi: 10.1097/IN9.0000000000000040. eCollection 2024 Apr. PMID 38680993

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03960333/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT03960333/ICF_001.pdf